CLINICAL TRIAL: NCT04545957
Title: Judging MR Simulation Procedures: A Phase I-II Study of the Use of Magnetic Resonance Imaging Simulation in the Planning of Radiation Treatments
Brief Title: Jump: MR Simulation For Radiation Therapy Master Protocol
Acronym: JUMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond Mak, Principal Investigator, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-759
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Recurrent Adenocarcinoma; Liver Cancer; Head and Neck Cancer
Keywords: Prostate Cancer; Recurrent Adenocarcinoma; Liver Cancer; Head and Neck Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Liver Neoplasms; Head and Neck Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Phase I MRI Simulation (Experimental): This research study involves a screening period to determine eligibility.
  - Radiation mapping to define the target for radiation.acquiring MR data at the specified timepoint in a patient's care plan and ability to identify the radiation target and develop a radiation therapy plan on the MR data.
  Interventions: Device: MRI Simulator; Radiation: Radiation Therapy
- Phase II MR Simulation Protocol: Track A (Experimental): MR-only Radiation Therapy Simulation MRI-simulation and synthetic CT to plan treatment
  Interventions: Device: MRI Simulator; Radiation: Radiation Therapy
- Phase II MR Simulation Protocol: Track B (Experimental): Adjusted Margin or / Dose Painted RT Based on Imaging of MR Simulator (e.g. biological imaging or higher resolution imaging)
  Interventions: Device: MRI Simulator; Radiation: Radiation Therapy

INTERVENTIONS:
Device: MRI Simulator — Radiation mapping to define the target for radiation.acquiring MR data at the specified timepoint in a patient's care plan and ability to identify the radiation target and develop a radiation therapy plan on the MR data.
Radiation: Radiation Therapy — In Phase I, radiation will be institutional standard per disease site. In Phase II, either radiation according to MR-based dose painting or adjusted RT. These adjusted doses and/or RT will vary per disease site and will be pre-specified in the subprotocols.

SUMMARY:
This is a master protocol for a prospective Phase I-II study evaluating feasibility and efficacy of incorporating magnetic resonance imaging (MRI) simulation into the planning of radiation treatments.

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. A Phase I clinical trial tests the feasibility and safety of an investigational intervention. "Investigational" means that the process targeting high doses of radiation to the tumor based on MRI is still being studied. This research study is a Feasibility Study, which means it is the first-time investigators at this institution are examining this type of MR-guided dose planning. The U.S. Food and Drug Administration (FDA) has cleared MRI planning for use.

* In Phase I of this study, will prospectively determine the feasibility of using an MRI simulator to plan radiation therapy.
* In Phase II, the efficacy of adjusting RT based on MRI simulation will be explored, either by utilizing an MRI-simulation and synthetic CT to plan treatment or by dose-painting based on functional MRI data

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed malignancy requiring radiation therapy.
* Age: 18 years or older
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Ability to understand and the willingness to sign a written informed consent document.
* Disease-specific eligibility criteria will be specified in the appropriate subprotocol.

Exclusion Criteria:

* For MRI involving contrast, history of allergic reactions attributed to gadolinium based IV contrast. Note: If patient will not receive contrast, this is not applicable
* Participants who cannot undergo an MRI
* Disease-specific exclusion criteria will be specified in the appropriate subprotocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2030-10-22 (Estimated); Study Completion 2030-10-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility of acquiring MRI simulation prior to radiation therapy planning | 1 Year
  Feasibility is defined as successfully enrolling patients, successfully acquiring MR data at the specified timepoint in a patient's care plan and ability to identify the radiation target and develop a radiation therapy plan on the MR data
Proportion of patients with QOL decline exceeding 2 x MID | baseline up to 24 months
  12 points; MID of the EPIC-26 urinary irritative/obstructive domain is 6 points) measured by EPIC-26 urinary irritation/obstruction domain from baseline to 2 years

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 24 Months
MRI evidence of disease at 2 years from treatment initiation. | 24 Months
PSA progression (nadir + 2) at 2 years from treatment initiation | 24 months
Progression free survival | 24 months
Change in target volumes between CT simulation and MRI simulation | 24 Months
  To ascertain the effects of MRI simulation on size of target volumes and OAR, the volume (cc) will be compared between CT vs MR simulation by t-test for normal data or Wilcoxon signed-rank test if data does not follow a normal distribution. The extent of overlap calculated with the Sorensen-Dice coefficient and Hausdorff distance.
Change in coverage of target volumes between CT simulation and MRI simulation | 24 Months
  The dose to OARS using the CT-simulation and MR-simulation derived plans will be compared using the t-test for normal data or Wilcoxon signed-rank test if data does not follow a normal distribution.
Change in dose to organs at risk (OARs) between CT simulation and MRI simulation | 24 Months
  The dose to OARS using the CT-simulation and MR-simulation derived plans will be compared using the t-test for normal data or Wilcoxon signed-rank test if data does not follow a normal distribution.
Performance of the synthetic CT in RT planning | 24 Months
  To assess performance of the synthetic CT in RT planning, fluence patterns from the synthetic CT plan will be copied onto the CT simulation electron density grids and dose recalculated. Accuracy of synthetic CT dose calculations to target volumes and OARs will be assessed with a goal of <1% difference in target and OAR dose between synthetic CT plans and CT simulation plans

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Mak, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation